CLINICAL TRIAL: NCT01115959
Title: Are Post Intracerebal Hemorrhage Prevented By Anti-Epileptic Treatment?
Brief Title: Seizures Post Intracerebral Hemorrhage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Yair Lampl, Professor Yair Lampl, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 001
Record Dates: First submitted 2010-05-02; First posted 2010-05-04 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2010-05

CONDITIONS: Post Cerebral Hemorrhage
MeSH Terms: interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- valproic acid (Active Comparator): Valproic acid given orally 400mg twice daily
  Interventions: Drug: valproic acid; Drug: placebo bid
- placebo (Placebo Comparator): Placebo twice daily for one month
  Interventions: Drug: placebo bid

INTERVENTIONS:
Drug: valproic acid — treatment of 1 month dosage of 400 mg BID
  Arms: valproic acid
Drug: placebo bid

SUMMARY:
This study examines early antiepileptic treatment with valproic acid for acute cerebral hemorrhage against a placebo group immediately post event to evaluate the outcome of these patients regarding seizures and neurological outcome.

ELIGIBILITY:
Inclusion Criteria:

* cerebral hemorrhage spontaneous

Exclusion Criteria:

* early seizures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2003-02; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
number of seizures | study drug for 1 month and 1 year follow up

SECONDARY OUTCOMES:
neurological outcome NIHSS | during 1 month study drug and 1 year post follow up

CONTACTS AND LOCATIONS:
Overall Officials: ronit gilad, md, Principal Investigator — E Wolfson med center; ronit gilad, md, Principal Investigator — E wofson med center